CLINICAL TRIAL: NCT04385199
Title: The Use of Convalescent Plasma for Patients Hospitalized With COVID-19 Disease
Brief Title: Convalescent Plasma for Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Geneva Tatem, Associate Clinical Professor of Medicine, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13807
Record Dates: First submitted 2020-05-09; First posted 2020-05-12 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Infection; Coronavirus; COVID
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma Intervention (Experimental): Convalescent plasma 200mL transfusion
  Interventions: Biological: Convalescent plasma
- Standard Therapy Control (No Intervention): Standard therapy for COVID-19 disease as defined by institutional protocols

INTERVENTIONS:
Biological: Convalescent plasma — One 200mL transfusion of ABO compatible convalescent plasma over 3 hours
  Arms: Convalescent Plasma Intervention

SUMMARY:
Pilot study of tolerability and efficacy of transfusion of 200mL of convalescent plasma in patients with COVID-19 respiratory disease.

DETAILED DESCRIPTION:
Importance: Convalescent plasma has been shown to be safe in patients with COVID-19, but whether it is clinically effective in patients with severe COVID-19 pneumonia is still unclear.

Objective: To evaluate the safety, tolerability, efficacy, and adverse events related to transfusion of convalescent plasma in patients hospitalized with severe or critical COVID-19 pneumonia.

Design, Setting and Participants: Randomized, single center, open-label, controlled trial of patients hospitalized between May 1, 2020, and August 1, 2020, with severe COVID-19 pneumonia in 1 tertiary care health system in the United States. A total of 30 participants age ≥ 18 years with 1 or more of the following were enrolled: dyspnea; respiratory rate > 30; O2 saturation ≤ 93%; PaO2/FiO2 or SaO2/FiO2 ratio < 300 mm Hg; and bilateral airspace opacities on chest x-ray > 50% within 24 to 48 hours.

Intervention: Transfusion with 1 unit of ABO compatible convalescent plasma in addition to standard care (n = 20) or standard care (n = 10). Standard care included steroids.

Main Outcomes and Measures: Primary outcome was improvement in oxygenation 72 hours after infusion measured by change in arterial blood gas or in PaO2/FiO2 or Sa/FiO2. Secondary outcomes were mortality at 28 days, days on mechanical ventilation, intensive care unit and hospital length of stay, and mSOFA score.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 with one or more of the following: Dyspnea Respiratory rate >= 30 breaths/min Oxygen saturation <=93% PaO2/FiO2 <300 Bilateral airspace opacities on chest radiograph at 24 to 48 hours

Exclusion Criteria:

* Acute myocardial infarction in past 30 days Acute stroke in past 30 days VV ECMO VA ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geneva Tatem, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Started | 20 | 10
Completed | 19 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 15 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.9) | 53 (13.6) | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity categories as defined by the National Institutes of Health/Office of Management and Budget (NIH/OMB) Standards
  Participants
    Hispanic or Latino | 3 | 5 | 8
    Not Hispanic or Latino | 13 | 3 | 16
    Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race categories as defined by the National Institutes of Health/Office of Management and Budget (NIH/OMB) Standards
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 13 | 3 | 16
    White | 3 | 5 | 8
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30
Dyspnea with Respiratory Rate (RR) >30 [Count of Participants; unit: Participants] — Number of participants with a respiratory rate >30 at randomization
  Participants | 9 | 4 | 13
SaO2/FiO2 [Mean (Standard Deviation); unit: ratio] — The ratio of oxygen saturation by pulse oximeter (SaO2) to oxygen concentration (FiO2)
  ratio | 188.4 (96.0) | 196.5 (89.9) | 190 (90)
Bilateral airspace opacities on CXR >50% within 24 to 48 hours [Count of Participants; unit: Participants] | 15 | 8 | 23
Mechanical ventilation [Count of Participants; unit: Participants] | 11 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Respiratory Disease Severity
Description: Change in oxygenation as documented by SaO2/FiO2 at 72 hours after infusion
Time Frame: day 3 post transfusion
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Number analyzed (Participants) | 20 | 10
ratio | 251 (89) | 276 (188)

2. Secondary Outcome: ICU Length of Stay
Description: Total ICU length of stay
Time Frame: Up to 60 days At the end of the trial, if patients were still in the ICU, their date of transfer out of the ICU was collected and total ICU length of stay calculated.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Number analyzed (Participants) | 20 | 10
days | 19.5 [10 to 46] | 13 [10 to 19]

3. Secondary Outcome: Length of Stay
Description: Hospital length of stay
Time Frame: Up to 60 days At the end of the trial, if patients were still in the hospital, their date of transfer out of the hospital was collected and hospital length of stay calculated.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Number analyzed (Participants) | 20 | 10
days | 20 [7.5 to 46] | 11.5 [9 to 18]

4. Secondary Outcome: Ventilator Days
Description: Duration of time on ventilator
Time Frame: 28 day
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Number analyzed (Participants) | 20 | 10
days | 15.6 [8.4 to 26] | 4.2 [1.4 to 7.5]

5. Secondary Outcome: Number of Participants With Transfusion Adverse Events
Description: Adverse transfusion events after 1 unit of convalescent plasma
Time Frame: From transfusion up to 1 day post-transfusion
Measure: Number; unit: participants
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Number analyzed (Participants) | 20 | 10
participants | 0 | 0

6. Secondary Outcome: Normal Chest X Ray at 28 Days
Description: Change in Chest X Ray Findings
Time Frame: 28 days
Population: Normal CXR at 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Number analyzed (Participants) | 20 | 10
Participants | 9 | 3

7. Secondary Outcome: All-cause Mortality
Description: All-cause overall deaths at end of trial at 28 days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma Intervention | Standard Therapy Control
Number analyzed (Participants) | 20 | 10
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 28 days
Groups:
- Intervention: Convalescent plasma 200mL transfusion
  Convalescent plasma: One 200mL transfusion of ABO compatible convalescent plasma over 3 hours
- Control: Standard therapy for COVID-19 disease as defined by institutional protocols
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 3/20 | 2/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04385199/Prot_SAP_000.pdf